CLINICAL TRIAL: NCT00757133
Title: Prevention of Incisional Hernia by Mesh Augmentation After Midline Laparotomy for Aortic Aneurysm Treatment.
Acronym: PRIMAAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008/379
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Conventional laparotomy closure
  Interventions: Procedure: Conventional laparotomy closure
- 2 (Active Comparator): Laparotomy closure with mesh augmentation
  Interventions: Procedure: Laparotomy closure with mesh augmentation

INTERVENTIONS:
Procedure: Conventional laparotomy closure — Recommended technique: The laparotomy is closed with a slowly resorbable running suture (f.e. PDS) in a single layer. The length of the suture should approximately be four (4) times the length of the fascial incision. The skin is closed with the usual technique of the department
  Arms: 1
Procedure: Laparotomy closure with mesh augmentation — Recommended technique: Mesh augmentation can be done in a retromuscular or a prefascial position. By consensus of the initial primary investigators a retromuscular (sublay) position of the mesh was chosen and as a mesh a light weight polypropylene mesh will be used. Retromuscular (sublay): (see reference no. 11: Rogers et al.) At the end of the vascular procedure the plane behind the rectus muscles (retromuscular-preperitoneal) is dissected as in a "Stoppa repair for incisional hernias"
  Arms: 2

SUMMARY:
The research hypothesis for this study is to possibly reduce the incidence of incisional hernia 2 years postoperatively after midline laparotomy for treatment of aortic aneurysm from 25% to 5% by mesh augmentation during closure of the laparotomy. The study is designed as a prospective randomised multi-centre trial, randomising patients in 2 groups concerning the surgical technique of the closure of the abdominal wall.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing elective Abdominal Aorta Aneurysm treatment through a midline laparotomy are eligible for the trial.
* All patients should sign the informed consent.

Exclusion Criteria:

* Patients below 18 years.
* Pregnancy.
* Emergency surgery for aortic aneurysm.
* Presence of mesh in the abdominal wall on the midline from previous operations ASA score 4 or more.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To reduce the incidence of incisional hernia 2 years postoperatively after midline laparotomy for treatment of aortic aneurysm from 25% to 5% by mesh augmentation during closure of the laparotomy Incidence of incisonal hernia | 2 years postoperatively

SECONDARY OUTCOMES:
Incidence of incisonal hernia | 1 year and 5 years after surgery
VAS scores of pain at rest | 12, 24, 48, 72, 96, 120 hours , 4 weeks and 3 months after surgery
Duration of surgery | After surgery
Occurrence of post-operative complications | After 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Berrevoet, MD, Principal Investigator — University Hospital, Ghent; Filip Muysoms, MD, Principal Investigator — AZ Maria Middelares Ghent
Locations (8):
- Belgium (8):
  - Stedelijk Ziekenhuis Aalst, Aalst
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Imelda Ziekenhuis, Bonheiden
  - AZ Maria Middelares Ghent, Ghent
  - University Hospital Ghent, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
  - CHU Sart Tilman, Liège
  - Sint Augustinus (GZA ziekenhuizen), Wilrijk

REFERENCES:
- [Derived] Muysoms FE, Detry O, Vierendeels T, Huyghe M, Miserez M, Ruppert M, Tollens T, Defraigne JO, Berrevoet F. Prevention of Incisional Hernias by Prophylactic Mesh-augmented Reinforcement of Midline Laparotomies for Abdominal Aortic Aneurysm Treatment: A Randomized Controlled Trial. Ann Surg. 2016 Apr;263(4):638-45. doi: 10.1097/SLA.0000000000001369. PMID 26943336
- See also: Website of the University Hospital Ghent — http://www.uzgent.be